CLINICAL TRIAL: NCT01392690
Title: Evaluation of a Primary Prevention Program for Anxiety Disorders Using Story Books
Acronym: TrucsDeDom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Quebec en Outaouais (Other)
Responsible Party: Regional Health Board of Quebec - Outaouais district, Original name of the organization: Régie Régionale de la Santé de l'Outaouais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RegieRegionale-07-2000-05; Les Trucs de Dominique (Other: Now named : Agence de Santé et des Services Sociaux)
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Anxiety
Keywords: No condition; Primary prevention; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting list control - no intervention (No Intervention): No intervention. After the post-test they were offered the prevention program.
- Dominique's handy tricks (Experimental): Children assisted to 10 workshops where they learned exercises to control their stress and anxiety.
  Interventions: Behavioral: Dominique's Handy Tricks

INTERVENTIONS:
Behavioral: Dominique's Handy Tricks — Children assisted to 10 workshops where they learned exercises to control their stress and anxiety.
  Arms: Dominique's handy tricks

SUMMARY:
The purpose of this study is to assess the impact of a primary prevention program for anxiety disorders.

This study was completed between 2000 and 2002, with the final report transmitted to the Quebec ministry of health in 2003.

DETAILED DESCRIPTION:
This study reports the results of a study evaluating a book-supported prevention program "Dominique's Handy Tricks" for anxiety disorders in children aged 9 to 12 years of age. This cognitive-behavioural program is delivered using a combination of story-based books and workshop sessions. The originality of the program comes from the use of story books that were not developed for anxiety management specifically. Every session is based on a story describing characters facing common stressors in childhood and how they managed to cope with their daily problems. In our randomized control trial with 46 children, participation in the program lead to a significant improvement in coping skills, self-efficacy, anxiety sensitivity, signs of anxiety and phobic avoidance. The theoretical and practical elements underlying the delivery of this primary prevention programs are described. It is suggested that such an approach, without any labelling specific to anxiety disorders, can be useful in universal primary prevention programs.

ELIGIBILITY:
Inclusion criteria:

* Recruitment for this study was open to every child in the school and was carried out with the help of staff from schools in Gatineau and Saint-André Avelin, Quebec.
* A total of 73 children aged between 9 and 12 years of age were screened.

Exclusion criteria:

Since the program does not target a clinical population, the following exclusion criteria were used:

* (1) a global score > 75 on the Child Behavior Checklist;
* (2) a score > 60 on the Screen for Child Anxiety Related Emotional Disorders (SCARED, child version);
* (3) outliers on outcome measures administered at pre-test; and
* (4) children who did not show up for the first workshop. The final enrolled study sample consisted of 59 children.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2000-03; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Change from pre-program on the Coping scale for children and youth | Pre (week 0), Post (week 10), F-up (6-months)
  Self-report questionnaire. Participants were assessed before implementing the prevention program (pre), after the program (week 10) and at the 6-month follow-up.

SECONDARY OUTCOMES:
Change from pre-program on the Childhood anxiety sensitivity index | Pre (week 0), Post (week 10), F-up (6-months)
  Self-report questionnaire. Self-report questionnaire. Participants were assessed before implementing the prevention program (pre), after the program (week 10) and at the 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Bouchard, Ph.D., Principal Investigator — Universite du Quebec en Outaouais
Locations (1):
- Universite du Quebec en Outaouais, Gatineau, Quebec, Canada

REFERENCES:
- [Result] Stéphane Bouchard, Jean Gervais, Nadia Gagnier. Évaluation d'un programme de prévention primaire des troubles d'anxiété pour les enfants de 9 à 12 ans : les trucs de Dominique. Rapport de recherche présenté à la Régie régionale de la santé et des services sociaux de l'Outaouais, Direction de la santé publique. 2003. Library number: J506 A58 B68.2003 ISBN 2-89251-157-7